CLINICAL TRIAL: NCT05084378
Title: Prospective Randomized Evaluation of Emerging Novel Treatments for Infection Prophylaxis in Total Joint Replacement: A Pilot Study
Brief Title: Evaluation of Emerging New Treatments for Infection Prevention in Total Joint Replacement
Acronym: PREVENT-IT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor
Organization: McMaster University (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: PREVENT-IT
Record Dates: First submitted 2021-08-22; First posted 2021-10-19 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Periprosthetic Joint Infection; Draining Wound
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The orthopaedic team (including the study coordinators) cannot be blinded to the treatment allocation as the solutions are visually distinguishable and these individuals need to lead the data collection at their clinical site. The participants, the Adjudication Committee Members, and the data analysts will be blinded to the study treatment. Participants may request to be unblinded following the completion of their 12-month visit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Povidone-iodine Lavage and Local Antibiotics (Experimental): 1 litre of 0.35% povidone-iodine lavage solution will be used. 2 grams of Vancomycin antibiotic powder will be applied to the deep joint (deep to fascia) following lavage solution and immediately prior to closure.
  Interventions: Drug: Povidone-Iodine Lavage Solution; Drug: Topical Antibiotic
- Chlorhexidine Lavage and Local Antibiotics (Experimental): 1 litre of 0.05% chlorhexidine lavage solution will be used. 2 grams of Vancomycin antibiotic powder will be applied to the deep joint (deep to fascia) following lavage solution and immediately prior to closure.
  Interventions: Drug: Chlorhexidine Lavage Solution; Drug: Topical Antibiotic
- Normal Saline Lavage and Local Antibiotics (Experimental): 1 litre of sterile isotonic saline solution will be used. 2 grams of Vancomycin antibiotic powder will be applied to the deep joint (deep to fascia) following lavage solution and immediately prior to closure.
  Interventions: Drug: Topical Antibiotic; Drug: Saline Lavage Solution
- Povidone-iodine Lavage Solution with no Local Antibiotics (Experimental): 1 litre of 0.35% povidone-iodine lavage solution will be used immediately prior to closure.
  Interventions: Drug: Povidone-Iodine Lavage Solution
- Chlorhexidine Lavage Solution with no Local Antibiotics (Experimental): 1 litre of 0.05% chlorhexidine lavage solution will be used immediately prior to closure.
  Interventions: Drug: Chlorhexidine Lavage Solution
- Normal Saline Lavage with no Local Antibiotics (Active Comparator): 1 litre of sterile isotonic saline solution will be used immediately prior to closure.
  Interventions: Drug: Saline Lavage Solution

INTERVENTIONS:
Drug: Povidone-Iodine Lavage Solution — 0.35% povidone-iodine solution mixed with 1 litre of sterile isotonic saline solution. Commercially available products with 0.35% povidone-iodine and sterile isotonic saline solution may also be used.
  Arms: Povidone-iodine Lavage Solution with no Local Antibiotics; Povidone-iodine Lavage and Local Antibiotics
Drug: Chlorhexidine Lavage Solution — 0.05% chlorhexidine solution mixed with 1 litre of sterile isotonic saline solution. Commercially available products with 0.05% chlorhexidine and sterile isotonic saline may also be used.
  Arms: Chlorhexidine Lavage Solution with no Local Antibiotics; Chlorhexidine Lavage and Local Antibiotics
Drug: Topical Antibiotic — 2 grams Vancomycin powder
  Arms: Chlorhexidine Lavage and Local Antibiotics; Normal Saline Lavage and Local Antibiotics; Povidone-iodine Lavage and Local Antibiotics
Drug: Saline Lavage Solution — 1 litre of sterile isotonic saline
  Arms: Normal Saline Lavage and Local Antibiotics; Normal Saline Lavage with no Local Antibiotics

SUMMARY:
At the end of total joint replacement (TJR) surgery, surgeons wash and clean the surgical wound. This is done to lower the risk of infections. Currently, most surgeons use saline to wash the surgical wound and do not place antibiotics in the wound . However, some recent studies have shown that using povidone-iodine and chlorhexidine-based solutions (both are types of antiseptics) to wash the surgical site and placing antibiotics directly into the wound may be effective in reducing infections in TJR surgery compared to saline and no antibiotics. However, no study has determined which solution is better at reducing the number of infections in patients undergoing TJR. The investigators also do not know if the addition of antibiotics applied to the wound will decrease infections. Currently, there are no surgical guidelines around infection prevention in total joint replacement. A large scale, multi-site, pragmatic 3 x 2 factorial randomized controlled trial is need that compares these six treatment groups. However, before this, a smaller pilot study must be conducted to determine the feasibility of a larger study. PREVENT-iT will address these important gaps in knowledge and clinical practice.

DETAILED DESCRIPTION:
The investigators propose a pilot study that will determine the feasibility of a definitive trial that compares irrigation fluids and topical antimicrobials to reduce the risk of wound complications requiring reoperation in patients undergoing primary or aseptic revision hip or knee TJR.

In the pilot phase, the investigators will compare three irrigation fluids (povidone-iodine lavage, chlorohexidine lavage, and normal saline) and the investigators will compare the use of vancomycin powder versus no powder in a 3 x 2 factorial RCT design.

Therefore, eligible and consenting participants will be randomized to one of six treatment groups:

1. Povidone-iodine lavage and local antibiotics
2. Chlorhexidine lavage and local antibiotics
3. Normal saline lavage and local antibiotics
4. Povidone-iodine lavage with no local antibiotics
5. Chlorhexidine lavage with no local antibiotics
6. Normal saline lavage with no local antibiotics

Study participants will be assessed at regular intervals in the one year following their TJR. The primary clinical outcome is PWD or PJI requiring reoperation within 90 days of TJR. The secondary clinical outcome is PJI within 12 months of TJR.

The time frame of 90 days was selected for the primary clinical endpoint (any reoperation for PWD or PJI) for the pilot phase of this study because the interventions may have a profound impact within the first three months after TJR. Measuring the primary outcomes at this time will allow the study team to examine any acute and early outcomes related to the intervention. This will also provide the study team with the opportunity to identify any potential problems with the interventions.

The one-year timeframe for the secondary clinical endpoint (PJI) was selected for the pilot phase of this study because the majority of PJIs are likely to be diagnosed with one year of TJR surgery. This time frame will allow the study team to record and analyze most of the PJIs, and like the primary outcomes, it will allow for the examination of early outcomes, and any potential problems with the treatments.

The investigators hypothesize the following:

1. Patients who have their surgical wound irrigated with either povidone-iodine or chlorhexidine will have a significantly lower rate of PWD and PJI requiring reoperation compared to patients who have their wound irrigated with saline.
2. Patients who have their surgical wound irrigated with povidone-iodine will have similar rates of PWD and PJI requiring reoperation as compared to patients treated with chlorohexidine.
3. Patients who receive topical vancomycin will have a significantly lower rate of PWD and PJI requiring reoperation compared to patients who did not receive topical antibiotics.
4. Patients who have their surgical wound irrigated with either povidone-iodine or chlorhexidine will have a significantly lower rate of PJI compared to patients who have their wound irrigated with saline.
5. Patients who have their surgical wound irrigated with povidone-iodine will have similar rates of PJI compared to patients treated with chlorohexidine.
6. Patients who receive topical vancomycin will have a significantly lower rate of PJIs compared to patients who did not receive topical antibiotics.

Participants will be followed for one year for safety and in anticipation that the pilot study may continue into the definitive trial phase. At the conclusion of the pilot study, the Principal Investigators will determine whether to:

* Continue with the existing protocol and proceed with the definitive trial.
* Revise the protocol based on lessons learned from the pilot phase.
* Conclude that the trial is not feasible.

The feasibility objectives in our pilot study do not lend themselves to traditional quantitative sample size calculations. The sample size for the pilot study will be 500 patients. This sample size for the pilot study was chosen in consideration of the following items:

* Due to the low event rate of PJI/PWD in this population, our initial sample size estimates suggest that the investigators will need a sample size of approximately 20,000 patients for the definitive trial. Given the large size of the definitive trial, a larger than usual sample size of 500 participants is needed and will represent approximately 2.5% of the sample size of a definitive trial. This will provide sufficient data to inform feasibility, sample size, and refine the design of the proposed definitive trial.
* As the definitive trial will have a large sample size and will be international in scale, the investigators need to demonstrate to our potential funding agencies our ability to enroll a high number of patients and maintain high level data collection and follow-up.
* The investigators also require a sufficient number of events in the pilot study to establish the adjudication process. A sample size of 500 participants will allow for the reporting and adjudication of approximately 15 events.

Statistical Methods:

Analysis Plan Overview The analysis and reporting of results will follow the CONSORT guidelines for reporting of randomized pilot and feasibility trials. The investigators will use descriptive statistics, reported as count and percentage or mean and standard deviation depending on the type of variable to summarize the results of our feasibility objectives of this pilot study. Feasibility outcomes will be based on descriptive statistics reported as % (95% CI).

The analyses will be conducted using R (Vienna, Austria).

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older.
2. Undergoing primary or revision TJR.
3. Informed consent obtained.

Exclusion Criteria:

1. Received antibiotics for any reason in the two weeks prior to their TJR.
2. Chronic or acute infection at or near the TJR site.
3. Prior history of PJI.
4. Undergoing surgery for a diagnosis of a fracture.
5. Open wounds on affected limb.
6. Undergoing bilateral TJR.
7. Medical contraindication to povidone-iodine.
8. Medical contraindication to chlorhexidine.
9. Medical contraindication to vancomycin.
10. Current or anticipated incarceration.
11. Terminal illness with expected survival less than 90 days.
12. Currently enrolled in a study that does not permit co-enrollment.
13. Unable to obtain informed consent due to language barriers.
14. Problems, in the judgment of study personnel, with maintaining follow-up with the patient.
15. Prior enrollment in the trial.
16. Other reason to exclude the patient, as approved by the Methods Centre.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2024-08-04 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Feasibility of a Definitive Trial based on the following criteria domains: 1) Participant Enrollment, 2) Administration of Treatments, 3) Data Collection Methods, and 4)Compliance with the Protocol. | 2 - 2.5 years
  Each domain will be interpreted via a "traffic light" approach, in which "green" will indicate moving forward as is with the definitive trial, "yellow" will mean proceeding with some modifications, and "red" will indicate that the definitive trial is not feasible. Feasibility criteria will be monitored over the course of the pilot study and modifications will be made to the protocol during the pilot phase to increase feasibility.

SECONDARY OUTCOMES:
Persistent Wound Drainage (PWD) and Periprosthetic Joint Infections (PJI) requiring reoperation | Within 90 days of the Total Joint Replacement Surgery
  Incidence of PWD and PJI events requiring reoperation will be measured. PWD will be defined as a non-infectious disturbance in wound healing of short duration that occurs during the days following TJR. PJI will be defined by the Musculoskeletal Infection Society (MSIS) criteria for diagnosis of PJI. Reoperations will include, but are not limited to, irrigation, debridement, liner exchange, and implant exchange. Reoperations for hardware complications or fracture will not be considered study events. A blinded Adjudication Committee will review all reported reoperations to confirm that they meet the criteria for being a study event.

OTHER OUTCOMES:
Tertiary/exploratory Outcome: Periprosthetic Joint Infections (PJI) | Within 12 months of the Total Joint Replacement Surgery
  Incidence of PJI events will be measured. PJI will be defined by the Musculoskeletal Infection Society (MSIS) criteria for diagnosis of PJI. Reoperations will include, but are not limited to, irrigation, debridement, liner exchange, and implant exchange. Reoperations for hardware complications or fracture will not be considered study events. A blinded Adjudication Committee will review all reported reoperations to confirm that they meet the criteria for being a study event.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wood, MD, Principal Investigator — McMaster University
Locations (6):
- Canada (4):
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Hamilton Health Sciences- Juravinkski Hospital, Hamilton, Ontario
  - Montreal General Hospital, Montreal, Quebec
  - St. Mary's Hospital, Montreal, Quebec
- Spain (2):
  - Hospital Clinic Barcelona, Barcelona
  - Vall d'Hebron University Hospital, Barcelona

IPD SHARING:
Plan to Share IPD: No